CLINICAL TRIAL: NCT05858606
Title: Pilot Study of Ethiology Research by a Multidisciplinary Evaluation Then a Genome-wide Analysis in a Cohort of Idiopathic Short Stature Patients
Brief Title: Multidisciplinary Evaluation and a Genome-wide Analysis in a Cohort of Idiopathic Short Stature Patients
Acronym: PAG PETI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL22_0396
Record Dates: First submitted 2023-04-07; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Idiopathic Short Stature
Keywords: idiopathic short stature; whole genome analysis; monogenic conditions; syndromic disorders; skeletal dysplasia
MeSH Terms: conditions — Mucopolysaccharidosis IV

STUDY DESIGN:
Intervention Model Description: Our trial aims to evaluate the prevalence of idiopathic short stature among children whose growth is above -2,5SD (AFPA- CRESS/Inserm -CompuGroup Medical 2018 curve) or above -2SD of the parental target size (taking child gender into account), after exclusion of classical pediatric and endocrinologic pathologies, and to evaluate the prevalence of monogenic causes of idiopathic short stature. We propose to perform a two-step study. The first one consists in a standardized multidisciplinary clinico-radiological evaluation of those children to evaluate the real prevalence of idiopathic short stature (ISS) among these patients. The second step consists in performing a whole genome sequencing analysis in the 30 first patients for whom the diagnosis of ISS is confirmed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 200 patients with idiopathic short stature, (Experimental): 200 patients with apparently idiopathic short stature,
  Interventions: Diagnostic Test: Evaluation of the prevalence of truly (authentified) idiopathic short stature after multidisciplinary clinico-radiological evaluation; Procedure: analysis in a multidisciplinary consultation meeting via a secure platform (ShareConfrère) for evaluation by multidisciplinary team; Genetic: Whole genome analysis for authentified idiopathic short stature

INTERVENTIONS:
Diagnostic Test: Evaluation of the prevalence of truly (authentified) idiopathic short stature after multidisciplinary clinico-radiological evaluation — 1. pre-inclusion consultation
  2. inclusion consultation
     * personal history
     * height, weight, cranial perimeters, and spans of both parents
     * clinical examination of the child
     * photographs of the child
     * additional X-rays
Procedure: analysis in a multidisciplinary consultation meeting via a secure platform (ShareConfrère) for evaluation by multidisciplinary team — multidisciplinary team (geneticist, orthopedist, radiologist, pediatric endocrinologist) which will assign each patient an orientation:
  * either to the non idiopathic short stature group (syndromic diagnostic orientation or to a constitutional bone pathology)
  * or to the authentified idiopathic short stature group
Genetic: Whole genome analysis for authentified idiopathic short stature — For the first 30 patients included in the authentified idiopathic short stature group, a whole genome analysis in trio (child + parents) will be performed as part of the research.
  For these 30 patients in the authentified idiopathic short stature group, the teleconsultation carried out for the submission of the multidisciplinary consultation meeting conclusions will make it possible to establish the family tree, to explain the interest and limits of the analysis, and to submit the consents dedicated to the genetic analysis.

SUMMARY:
Our trial aims to evaluate the prevalence of idiopathic short stature among children whose growth is above -2,5SD (AFPA- CRESS/Inserm -CompuGroup Medical 2018 curve) or above -2SD of the parental target size (taking child gender into account), after exclusion of classical pediatric and endocrinologic pathologies, and to evaluate the prevalence of monogenic causes of idiopathic short stature. We propose to perform a two-step study. The first one consists in a standardized multidisciplinary clinico-radiological evaluation of those children to evaluate the real prevalence of idiopathic short stature (ISS) among these patients. The second step consists in performing a whole genome sequencing analysis in the 30 first patients for whom the diagnosis of ISS is confirmed.

DETAILED DESCRIPTION:
Detailed description: Establishing the etiological diagnosis of short stature is an important step to guide the therapeutic management of patients and to propose appropriate genetic counseling. Short stature can be a symptom of many pathologies. However, in the majority of cases (80%), no specific etiology is found during a pediatric clinical investigation. In this case, the diagnosis of "idiopathic" short stature is performed. However, the diagnostic and therapeutic management of short stature after exclusion of classical pediatric causes is extremely heterogeneous and there are currently no consensual recommendations. We could therefore expect to have a much higher proportion of diagnosed patients with more standardized procedures both clinical and genetic. Additionally, in recent years, new methods of genetic investigation (gene panel, whole exome or whole genome sequencing analysis) have made it possible to identify many genetic variants associated with apparently isolated short stature. So far, none of the publications reporting next-generation sequencing analysis have focused on patients with authentic idiopathic short stature, i.e. without associated bone anomalies or syndromic features, and are often focused on only a subset of target genes.

Our trial aims at estimating the prevalence of idiopathic short stature among children whose growth is above -2,5SD (AFPA- CRESS/Inserm -CompuGroup Medical 2018 curve) or above -2SD of the parental target size, after exclusion of classical pediatric and endocrinologic pathologies, and to evaluate the prevalence of monogenic causes of idiopathic short stature. We propose to perform a two-step study. The first one consists in a multidisciplinary clinico-radiological evaluation of those children to evaluate the real prevalence of idiopathic short stature (ISS) among these patients. The second step consists in performing a whole genome sequencing analysis in the 30 first patients for whom the diagnosis of authentic ISS is confirmed.

All patients will have:

* a pre-inclusion visit
* an inclusion visit after which the multidisciplinary clinico-radiological evaluation will be held

This analysis will assign patients to the diagnosis of either:

1. non-idiopathic short stature (diagnosis of constitutional bone disease or syndromic disorder)
2. authentic idiopathic short stature

A teleconsultation (1) to explain to the parents the conclusions of the multidisciplinary clinico-radiological evaluation.

This teleconsultation will be followed for all patients in the "non-idiopathic short stature" group, by a visit to take samples for genetic analysis in the context of clinical care, followed by a teleconsultation (2) to give them and explain the results

This teleconsultation will be followed for the first 30 patients in the "authentified idiopathic short stature" group, by a visit to take samples for whole genome analysis in the context of research, followed by a teleconsultation (2) to return the results.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4 to 18 years
* 2 sexes
* Height less than -2.5DS (standard deviations of the AFPA- CRESS/Inserm -CompuGroup Medical 2018 curve) or less than -2DS of the TCP (parental target height, corresponding to the average of parental heights +6.5 cm in boys, -6.5 cm in girls)
* Normal karyotype + FISH SHOX for girls
* Previously performed:celiac disease antibodies, WBC-platelets, CRP, blood ionogram, creatinine, blood calcium, blood phosphorus, ASAT, ALAT, PAL, PTH, TSH, T4L, growth hormone test normal according to the standards of the laboratory of the CHU of Montpellier
* Acceptance of X-rays, in addition to those already performed as part of the care, which will not be repeated if necessary: spine front and profile, pelvis front, 1 upper limb front, 1 lower limb front F, hands and feet front
* Acceptance of photographs: whole body with underwear, face face and profile, 2 faces of hands; feet, face
* Acceptance of blood samples for the child and the 2 parents (trio)
* Consent signed by both parents

Exclusion Criteria:

* Intellectual disability (IQ below 70)
* Cardiac, renal, digestive or cerebral malformation, cleft lip or palate, hearing or visual impairment, epilepsy
* Renal or cardiac insufficiency, digestive or chronic inflammatory pathology
* Previously established genetic diagnosis

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
proportion of patients with authentified idiopathic short stature after multidisciplinary clinical-radiological analysis | 3 years
  Primary endpoint:
  The primary outcome is the proportion of patients with authentified idiopathic short stature after multidisciplinary clinical-radiological analysis (including geneticist, orthopedist, pediatric endocrinologist, radiologist) performed during a dedicated Multidisciplinary Consultation Meeting (MCM)

SECONDARY OUTCOMES:
Genome positivity rate | 3 years
  Genome positivity rate (positive diagnosis of pathogenic variation (class 5, Figure 3) or probably pathogenic variation (class 4, Figure 3) variants involved in the phenotype) in the group of 30 patients with authentified idiopathic short stature patients in whom the genome analysis was performed
Rate of positivity of molecular analyses prescribed as part of the care following the PCR | 3 years
  Rate of positivity of molecular analyses prescribed as part of the care following the PCR (positive diagnosis of pathogenic or probably pathogenic variants involved in the phenotype) for patients with non-idiopathic short stature
Rate of modification of management by the results of genome analysis | 3 years
  Rate of modification of management by the results of genome analysis in the group of 30 patients with authentified idiopathic short stature in whom genome analysis has been performed
Type of change in management due to genome analysis results | 3 years
  Type of change in management due to genome analysis results: initiation/withdrawal of treatment, referral to organ specialist for specific multidisciplinary management (patients with authentified idiopathic short stature/ Genome+)
Rate of change in management by results of molecular analysis performed in a patient-care context for those with non-idiopathic short stature | 3 years
Type of management modification by molecular analysis resultscare context for those with non-idiopathic short stature | 3 years
  Type of management modification by molecular analysis results: initiation/withdrawal of treatment, referral to organ specialist for specific multidisciplinary management (patients with non-idiopathic short stature).
Parental satisfaction assessed via a visual analog scale (Teleconsultation (1) and (2)) | 3 years
Variants within the same gene identified in at least 2 patients by whole genome analysis in the group of 30 patients with authentified idiopathic short stature in whom genome analysis has been performed | 3 years